CLINICAL TRIAL: NCT06507943
Title: Community Health Equity Accelerator (CHEA): Community-Academic Asthma Partnership, Pediatric Asthma Intervention
Brief Title: Community Health Equity Accelerator (CHEA) Pediatric Asthma Intervention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Hispanic Federation, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2000037314
Record Dates: First submitted 2024-07-11; First posted 2024-07-18 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Asthma in Children
Keywords: Medical Legal Partnership; Community Health Worker; Health Harming Legal Needs

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Promotora (Experimental): Two Hispanic Federation Promotoras (community health workers) will provide culturally competent, bilingual home visits for asthma-related education and evaluation and support for health-harming legal needs (e.g., mold, rodents), including an initial visit and a follow-up visit 6-8 weeks later.
  Interventions: Behavioral: Promotora Home Visit

INTERVENTIONS:
Behavioral: Promotora Home Visit — For each participating family, Promotora home visits will be scheduled 6-8 weeks apart, with in-person or virtual visits conducted per the family's preference. The visits will begin with a survey which will evaluate concerns related to asthma for the child and the family, including their asthma control (via the ACT), their home environment (via screening for environmental exposures), and quality of life for the child. These surveys will be available in both online or physical forms for potential connectivity concerns, and Promotoras will have IPads for the online forms. The Promotoras, who have received specialized asthma training, will then address concerns raised by families, using the Clinical Pathway which will have resources for asthma-related concerns that are raised.

SUMMARY:
The purpose of this pilot is to initiate an academic-community partnership and launch a multi-level intervention that includes an asthma exposure pathway (an online decision support and resource) and a health Promotora program that will provide culturally responsive asthma support alongside legal and medical services to improve access to asthma care and ultimately improve asthma-related outcomes in the New Haven region.

DETAILED DESCRIPTION:
In this will be a prospective, non-randomized, observational, multi-level pilot intervention, general pediatricians and specialists in New Haven, Connecticut will utilize a newly developed clinical pathway that will be publicly available at the Yale Pediatrics Clinical Pathways website and accessible within the electronic health record (EHR) via integrated software to submit referrals for participants in a Promotora (Community Health Worker) asthma home-visiting intervention.

The Hispanic Federation Promotoras, who are partners in this study who have received Human Subjects research training, will enroll participants in the study. For each participating family, Promotora home visits will be scheduled 6-8 weeks apart, with in-person or virtual visits conducted per the family's preference. The Promotoras, who have received specialized asthma training, will address concerns raised by families, using the clinical pathway as a resource (the pathway will have resources for asthma-related concerns that are raised). A clinician from the study team will be on call at all times for the Promotoras in case urgent questions arise, and weekly case-conferences will be arranged to discuss any additional needs for support.

In this study, the primary outcomes will include measures of feasibility of both Promotora home visits and pathway utilization. The investigators will evaluate secondary outcomes using an interrupted time series analysis to evaluate asthma-related outcomes. In addition to survey data, asthma exacerbation metrics will be collected from the electronic health record.

ELIGIBILITY:
Inclusion Criteria:

Children with a diagnosis of asthma with at least one of the following:

* Oral steroid prescription in past 12m
* ED visit for asthma in past 12m
* Hospital admission for asthma in past 12m
* Asthma control test (ACT) score at visit ≤19
* Concern for asthmogenic exposure in the home (such as mold, pests, smoking, or pollution)
* At least one missed follow-up appointment for asthma
* At least one asthma exacerbation in the prior year
* Interested in asthma education (such as education in how to prevent asthma or how to administer medications)
* Concern for medication non-adherence

Exclusion Criteria:

* Living outside of New Haven Zip Code

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Referrals Resulting in Home Visit, to Assess Feasibility of Promotora Visits | One Year
  Percent of referred participants (from all referrals placed) to the newly-established asthma home visiting Promotora Program that resulted in a home visit (in-person or virtual)
Percent of clinicians who use pathway, to assess feasibility of asthma pathway use | One Year
  Percent of clinicians at participating practices who have accessed the asthma intervention pathway (using data from pathway utilization metrics)
Percent of patients for whom the pathway is used, to assess feasibility of asthma pathway use | One Year
  Percent of patients for whom a clinician accessed the asthma pathway (using pathway utilization metrics) out of total potential children for whom it could be used (using deidentified electronic health (EHR) record data tool)
Count of use of individual asthma pathway component use | One Year
  Count of use of individual asthma pathway components (using pathway utilization metrics)

SECONDARY OUTCOMES:
Mean Asthma Control Test (ACT) for 4-11 years scores | Baseline and 6-8 weeks later
  The ACT (for 4-11 years) is a seven-item survey with likert scales for caregivers (3 questions, scores 0-5) and children (5 questions, scores 0-3) together. It is used to evaluate asthma control with total score range of 0 (poorly controlled) to 27 (well-controlled)
Mean Pediatric Quality of Life (Peds-QL) scores | Baseline and 6-8 weeks later
  The Peds-QL is a 15 item survey with likert scales (0-4), with transformed scores out of 100, with a score range of 0 (poor quality of life) to 100 (high quality life).
Mean number of hospital admissions for asthma | Two years (year before and year after intervention)
  Total number of hospital admissions for asthma, evaluated via manual count via chart review.
Mean number of emergency department (ED) visits for asthma | Two years (year before and year after intervention)
  Total number of ED visits for asthma, evaluated via manual count via chart review.
Mean number of urgent visits for asthma | Two years (year before and year after intervention)
  Total number of urgent visits for asthma, evaluated via manual count via chart review.
Mean number of oral steroid prescriptions for asthma | Two years (year before and year after intervention)
  Total number of oral steroid prescriptions for asthma, evaluated via manual count via chart review.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Rosenberg, MD MHS, Principal Investigator — Yale University
Locations (1):
- Yale, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No